CLINICAL TRIAL: NCT05854628
Title: The Role of Red Flavonoid in Photoaging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We decided not to proceed further to enroll patients.
Sponsor: Johns Hopkins University (Other)
Collaborators: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00384338
Record Dates: First submitted 2023-04-12; First posted 2023-05-11 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Photoaging of Skin; Skin Aging

STUDY DESIGN:
Intervention Model Description: Investigators will recruit up to 75 participants for the entire study. Approximately half will be randomly assigned to treatment group and half randomly assigned to placebo group. The treatment group participants will be given 0.1% red flavonoids facial cream while the control cohort will be given a placebo facial cream.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double blind, neither the participants nor the investigators will be aware of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.1% red flavonoids facial cream (Experimental): 0.1% red flavonoids facial cream
  Interventions: Procedure: skin biopsy
- Placebo facial cream (Placebo Comparator): Placebo moisturizing facial cream
  Interventions: Procedure: skin biopsy

INTERVENTIONS:
Procedure: skin biopsy — Skin biopsies will be obtained at different time points.

SUMMARY:
The goal of this clinical trial is to learn about the effects of "red flavonoid" substance on skin, which is extracted from a plant called Camellia japonica, in adults aged of 45 or older with photo-damaged skin.

The main questions it aims to answer are:

* Does red flavonoid have an anti-aging effect?
* Does red flavonoid have any skin quality-improving effects? Participants will
* Be using creams with or without red flavonoid (only moisturizing creams) and sun-screen for the duration of the study.
* Get a skin biopsy before and after using the creams.
* Be taken photos of the face and neck region and have a skin examination at each visit.
* Complete a self-questionnaire at final visit. Researchers will compare the group who uses red flavonoid facial cream with the group who uses moisturizing cream to see if red flavonoid has an effect on appearance and structure.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the anti-photoaging effects of red flavonoid, a product with natural phytochemical kaempferol tetrasaccharides (KTs) extracted from Camellia japonica. The investigators hypothesize that Red flavonoids extracted from Camellia japonica will present anti-aging effects, such as skin smoothening, increased elasticity, and brightening, with high subjective participant satisfaction and microscopically corroborating analyses.

Individuals will be recruited from patient populations seen at the general dermatology clinics of Johns Hopkins Department of Dermatology or from patient populations participating in Johns Hopkins Cutaneous Translational Research Program (CTReP) research studies. Study procedures will be conducted at the Johns Hopkins CTReP office located at the Johns Hopkins Outpatient Center. Once eligibility has been demonstrated, the potential subjects will be instructed to make the first study appointment. This feasibility study will have a study population of up to 75 individuals over the age of 45. Each study participant will have up to 7 on-site visits within 24 weeks. A facial cream with or without 0.1% red flavonoid will be provided for twice-daily use. At various time points, photographs and clinical assessments will be collected as well as punch biopsy samples for laboratory study.

At the discretion of the principal investigator, biopsies may be taken from subjects before and following daily usage of the product of interest, up to 8 biopsies in total. The timepoints may be adjusted as data is being collected. A punch biopsy procedure will be employed which is a routine dermatological procedure consisting of local anesthesia, followed by the punch, which cuts a cylindrical core of epidermis, dermis, and subcutaneous tissue. A biopsy size of up to 4-mm in diameter is considered enough to perform all tests required by this protocol. After removal of the tissue sample, a suture is placed to close the circular opening. Sutures are removed and a scar is formed, but typically heals well without complications and blends well with the surrounding skin.

Standardized digital photographs will be obtained by study staff using a digital camera and software under standard photographic conditions at each study visit. Participants' eyes will be blacked out to de-identify photos. Photograph files will be coded to remove personal identifiers and stored on a secure hard drive in CTReP.

Non-invasive clinical assessments will be performed to 1) record skin findings using graded scales if needed, 2) to identify suitable areas for biopsy, 3) give information/demonstration about the product of interest, 4) to identify occurrence of any adverse events and 5) record post treatment findings.

Tissue work-up may include, but not limited to hematoxylin and eosin staining for assessment of epidermal/dermal thickness, reverse transcription-polymerase chain reaction and immunohistochemistry for photoaging and pigmentation markers such as fibrillin-1, collagen type IV, or collagen type I, and tyrosinase.

Any clinical findings determined by the Investigator to be important and/or unusual will be referred to as an adverse event. Study participants are asked to contact clinic staff immediately if the participants experience a reaction to the topical applications at any time during the study. Expected reactions may be documented in a problem events log. The investigator will use his discretion to remove participants from the study, and all problem events will be reported to Institutional Review Board.

Differences in protein expression between the test sites, and after application of test substances for varying periods of time, will be assessed for significance using either Student's t-test or analysis of variance (or non-parametric equivalents, if necessary) depending on the comparison required.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe photo-aged skin that is within the Fitzpatrick skin types 1-6
* Must be healthy enough to undergo skin biopsy in the opinion of the investigator
* Must be willing to comply with the requirements of the protocol
* Must have the ability to understand and communicate with the investigator
* Must be able to provide informed consent.

Exclusion Criteria:

* Subjects who are unable to provide informed consent
* Subjects with history of keloid scars
* Subject with significant medical history or current skin diseases that the investigator feels is not safe study participation
* Subjects who have used products containing salicylic acid, beta hydroxyl acids or vitamins A, C, or E in the last 14 days
* Subjects who have used topical antibiotics or topical retinoids in the last 30 days
* Subjects who have had a recent surgical or esthetic procedure in the last 3 months that can affect facial wrinkles or facial hyperpigmentation, such as botulinum toxin injections, chemical peels, laser-based therapies to the face, or face lift surgeries
* Subjects with allergies to lidocaine or epinephrine
* Subjects who self-report as nursing/pregnant or planning to be pregnant during the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Fibrillin-1 fold change as determined by Reverse Transcription Polymerase Chain Reaction (RT-PCR) | 8 weeks, 16 weeks, 24 weeks
  The investigators will detect the fold change of Fibrillin-1 in the basal layer of the epidermis in both skin treated with Red Flavonoids and placebo, by RT-PCR, to determine whether Red Flavonoids can improve skin photodamage and aging.
Collagen type-4 fold change as determined by Reverse Transcription Polymerase Chain Reaction (RT-PCR) | 8 weeks, 16 weeks, 24 weeks
  The investigators will detect the fold change of Collagen type-4 in the basal layer of the epidermis in both skin treated with Red Flavonoids and placebo, by RT-PCR, to determine whether Red Flavonoids can improve skin photodamage and aging.
Collagen type-1 fold change as determined by Reverse Transcription Polymerase Chain Reaction (RT-PCR) | 8 weeks, 16 weeks, 24 weeks
  The investigators will detect the fold change of Collagen type-1 in the basal layer of the epidermis in both skin treated with Red Flavonoids and placebo, by RT-PCR, to determine whether Red Flavonoids can improve skin photodamage and aging.
Tyrosinase fold change as determined by Reverse Transcription Polymerase Chain Reaction (RT-PCR) | 8 weeks, 16 weeks, 24 weeks
  The investigators will detect the fold change of Tyrosinase in the basal layer of the epidermis in both skin treated with Red Flavonoids and placebo, by RT-PCR, to determine whether Red Flavonoids can improve skin photodamage and aging.
Wrinkles/photoaging as assessed by clinical assessments | 8 weeks, 16 weeks, 24 weeks
  Griffith's photonumeric scale will be used. It is a nine-point scale where 0 (zero) is no wrinkles/photodamage and 8 is severe wrinkles/photodamage.
Hydration as assessed by clinical assessments | 8 weeks, 16 weeks, 24 weeks
  Skin hydration will be graded with a five-point scale where 0 (zero) is adequate hydration and 4 is severe dehydration.
Loss of elasticity as assessed by clinical assessments | 8 weeks, 16 weeks, 24 weeks
  Loss of elasticity will be graded as absent, localized or diffuse.
Brightness as assessed by clinical assessments | 8 weeks, 16 weeks, 24 weeks
  Brightness improvement rate will be graded with a five-point scale where 0 (zero) is marked improvement and 4 is no improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chien, MD, Principal Investigator — Johns Hopkins School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pereira AG, Garcia-Perez P, Cassani L, Chamorro F, Cao H, Barba FJ, Simal-Gandara J, Prieto MA. Camellia japonica: A phytochemical perspective and current applications facing its industrial exploitation. Food Chem X. 2022 Feb 17;13:100258. doi: 10.1016/j.fochx.2022.100258. eCollection 2022 Mar 30. PMID 35499017
- [Result] An S, Cho SY, Kang J, Lee S, Kim HS, Min DJ, Son E, Cho KH. Inhibition of 3-phosphoinositide-dependent protein kinase 1 (PDK1) can revert cellular senescence in human dermal fibroblasts. Proc Natl Acad Sci U S A. 2020 Dec 8;117(49):31535-31546. doi: 10.1073/pnas.1920338117. Epub 2020 Nov 23. PMID 33229519
- [Result] Kim J, Kim HS, Choi DH, Choi J, Cho SY, Kim SH, Baek HS, Yoon KD, Son SW, Son ED, Hong YD, Ko J, Cho SY, Park WS. Kaempferol tetrasaccharides restore skin atrophy via PDK1 inhibition in human skin cells and tissues: Bench and clinical studies. Biomed Pharmacother. 2022 Dec;156:113864. doi: 10.1016/j.biopha.2022.113864. Epub 2022 Oct 14. PMID 36252351
- [Result] Mukherjee S, Date A, Patravale V, Korting HC, Roeder A, Weindl G. Retinoids in the treatment of skin aging: an overview of clinical efficacy and safety. Clin Interv Aging. 2006;1(4):327-48. doi: 10.2147/ciia.2006.1.4.327. PMID 18046911
- [Result] Sitohang IBS, Makes WI, Sandora N, Suryanegara J. Topical tretinoin for treating photoaging: A systematic review of randomized controlled trials. Int J Womens Dermatol. 2022 Mar 25;8(1):e003. doi: 10.1097/JW9.0000000000000003. eCollection 2022 Mar. PMID 35620028